CLINICAL TRIAL: NCT05193266
Title: Gastroesophageal Reflux Disease and Its Health-related Quality of Life Among ICU Survivors
Brief Title: Gastroesophageal Reflux Disease (GERD) Among ICU Survivors
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Professor, Critical Care Medicine, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2021-265-DM-EXP-43
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Gastroesophageal Reflux Disease; Critically Ill
Keywords: Gatroesophageal reflux disease; Critically ill; Health-related quality of life; Outcome; Survivors; Intensive care unit
MeSH Terms: conditions — Gastroesophageal Reflux; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
Gastro-esophageal reflux disease (GERD) is a condition characterized by reflux of stomach contents causing troublesome symptoms and complications. Typical symptoms include heart burn (a retrosternal burning sensation), regurgitation (perception of flow of refluxed stomach content into the mouth or hypopharynx) and chest pain. As per recently published global guidelines (2017) by World Gastroenterology Organisation (WGO), the presence of heartburn and/or regurgitation symptoms 2 or more times a week is suggestive of GERD. Global burden of GERD in general population is approximately 1.03 billion, the prevalence of GERD varies geographically, with the highest prevalence of 19.55% in North America while in Asia, the estimated rate is 12.92%. However the data regarding the prevalence of GERD in intensive care unit (ICU) population is not yet established; which is expected higher after recovery from their current acute illness. In a healthy individual, several factors contribute to the prevention of reflux and to minimizing esophageal acid exposure: lower esophageal sphincter (LES) pressure, the diaphragmatic crura, gravity, esophageal peristalsis, salivary bicarbonate and the integrity of esophageal epithelium. But in critically ill these factors are compromised leading to high incidence of GERD. Interventions commonly used in managing critically ill patients such as sedation, presence of an endotracheal tube, mechanical ventilation, enteral tube feedings, positioning, and medications, along with specific patient characteristics and comorbid conditions contribute to an increased risk for GERD in this population. GERD results in various symptoms which has impact on quality of life. Various reliable and validated generic and disease specific instruments are available to measure symptom severity of the disease. In the present study, among GERD patients, commonly and freely available GERD-Health-related quality of life (GERD-HRQL) score will be used which is a disease-specific instrument. This observational study will screen and enroll adult patients who survived at the time of ICU discharge.

DETAILED DESCRIPTION:
During study period, all patients who survived at the time of ICU discharge will be considered as per inclusion and exclusion criteria. All eligible participants will be screened for the presence of GERD. If GERD present, participants will be followed for their symptoms after 6 week of the ICU discharge. Participant who did not having GERD at the time of ICU discharge will also be followed for the presence of GERD symptoms at 6 weeks after ICU discharge, if participant develop GERD symptoms then they will be followed up again for next 6 weeks. In participants who had GERD symptoms, HRQL score will be collected including 6-week follow up, after obtaining the informed written consent.

Demographic and clinical characteristics of all eligible participants will be collected on structured proforma. ICU prognostication scores, i.e., Acute Physiologic and Chronic Health Evaluation (APACHE) II score and Sequential Organ Dysfunction Assessment (SOFA) will be noted. All relevant and possible risk factors during ICU stay will also be collected. Participants with GERD, GERD-HRQL score will be collected, including 6-week follow-up.

At the time of ICU discharge, participant will be asked for the preference for the way of communication during follow-up with the option of pre-stamped envelope for postal with questionnaire. Participants will be handed over these envelopes with mention of pre-defined follow-up date for that particular patient. In case participant has plan for SGPGIMS visit for his/her pre-scheduled follow-up with any specialty, then data for present study will be collected in person.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) who survived at the time of ICU discharge

Exclusion Criteria:

* ICU stay <96 hours
* At the time of ICU discharge GCS <15
* Presence of open abdomen (post surgery)
* Presence of feeding tube at the time of ICU discharge
* Presence of abdominal drain or PEG tube at the time of ICU discharge
* Presence of tracheostomy tube at the time of ICU discharge
* Patient who do not provide written consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critically ill adult patients who survived at the time of ICU discharge
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of Gatroesophageal reflux disease (GERD) among ICU survivors | 12 weeks after ICU discharge
  Percentage of ICU survivors among whom Gatroesophageal reflux disease (GERD) present

SECONDARY OUTCOMES:
Gatroesophageal reflux disease-Health-related quality of life score among GERD present patients | 12 weeks after ICU discharge
  Gatroesophageal reflux disease-Health-related quality of life score will be measured two times (6 weeks apart). The minimum score is 0 and maximum score is 50. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Department of Critical Care Medicine, Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh, India